CLINICAL TRIAL: NCT02554409
Title: Sanofi Pasteur Quadrivalent Intradermal Influenza Vaccine Pregnancy Registry Protocol
Brief Title: Sanofi Pasteur Quadrivalent Intradermal Influenza Vaccine Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: QID02; U1111-1161-3485 (Other: WHO)
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy; Influenza
Keywords: Fluzone Quadrivalent Intradermal Influenza Vaccine; Pregnancy Registry; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnancy Cases: No Intervention as part of this protocol
  Interventions: Biological: Quadrivalent Intradermal Influenza Vaccine (QIV)

INTERVENTIONS:
Biological: Quadrivalent Intradermal Influenza Vaccine (QIV) — No Intervention as part of this protocol

SUMMARY:
The Sanofi Pasteur Fluzone Intradermal Quadrivalent vaccine (Fluzone QIV-ID) Pregnancy Registry will be a prospectively recruited pregnancy surveillance program designed to collect to collect and analyze information on vaccine exposures, pregnancy outcomes, and fetal and offspring outcomes on pregnant women exposed to Fluzone QIV-ID vaccine.

DETAILED DESCRIPTION:
Sanofi Pasteur will encourage registration of pregnant women exposed to Fluzone QIV-ID in the Sanofi Pasteur Pregnancy Registry by providing the registry's toll-free number, 1-800-VACCINE (1-800-822-2463), in the USPI. The toll-free number will also be available through the Sanofi Pasteur-sponsored Website for the Pregnancy Registry. Both the United States product insert (USPI) and Website will advise health care providers to register women who are pregnant or became aware they were pregnant at the time of Fluzone QIV-ID immunization.

Descriptive statistical methods will be the primary approach for summarizing data from the Fluzone QIV-ID Pregnancy Registry. No vaccine products will be provided or administered as part of this registry protocol.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women will be enrolled in the registry prospectively (after exposure to a product but before the conduct of any prenatal tests that could provide knowledge of the outcome of pregnancy). If the condition of the fetus has already been assessed through prenatal testing (e.g., targeted ultrasound, amniocentesis, etc.), such reports will be considered retrospective reports. Retrospective reports are also eligible for the registry, but they will be analyzed separately from prospective reports.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women exposed to Sanofi Pasteur's Quadrivalent Intradermal Influenza Vaccine (QIV ID)
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Number of cases and outcomes of pregnancies following exposure to QIV ID vaccine. | Up to six years
  Data will be summarized using descriptive statistical methods and stratified by pregnancy outcome (spontaneous abortion, elective termination, fetal death stillbirth, live birth) and timing of vaccine exposure. Infant outcomes include birth defects and physical and social development.

CONTACTS AND LOCATIONS:
Overall Officials: Product Safety Officer, Study Director — Sanofi Pasteur Inc.
Locations (5):
- United States (5):
  - San Diego, California
  - Miami, Florida
  - Albany, New York
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com
- See also: Sanofi Pasteur Pregnancy Registry — http://www.sanofipasteurpregnancyregistry.com/